CLINICAL TRIAL: NCT03772951
Title: The Efficacy for Execution Function and Genetic Mechanism of Computerized Cognitive Remediation Therapy for Chronic Schizophrenia
Brief Title: The Efficacy of Computerized Cognitive Remediation Therapy for Chronic Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKQ201813
Record Dates: First submitted 2018-10-24; First posted 2018-12-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation Therapy (Active Comparator): The study group received antipsychotic drugs Clozapine combined with Computerized Cognitive Remediation Therapy for 4 times/week for 45 minutes each time. For a total of 12 weeks. Clozapine, dosage, dosage form, and frequency :300~600 mg/d; po; duration: 12 week.
  Interventions: Other: Cognitive Remediation Therapy; Drug: Clozapine
- Clozapine (Placebo Comparator): Clozapine, dosage, dosage form, and frequency :300~600 mg/d; po; duration: 12 week.
  Interventions: Drug: Clozapine

INTERVENTIONS:
Other: Cognitive Remediation Therapy — Through computer information technology, using error-free, procedural learning, speech enhancement and a series of targeted computer programmatic cognitive correction tasks, patients can gradually improve problem solving and information processing capabilities, thereby improving their recognition function.
  Other Names: CCRT
  Arms: Cognitive Remediation Therapy
Drug: Clozapine — the course of disease is more than 2 years, the condition is stable for more than one month
  Other Names: CLZ

SUMMARY:
The study group received antipsychotic drugs combined with Computerized Cognitive Remediation Therapy (CCRT) for 4 times/week for 45 minutes each time. The control group only received antipsychotic drugs. For a total of 12 weeks. Brain Derived Neurotrophic Factor (BDNF) and Tropomyosin-related kinase B (Trk B) genes in peripheral blood were detected in both groups before and after treatment. Clinical symptoms and executive function assessment were performed in both groups before and after treatment. The relevance of genes and their effects on downstream protein expression levels led to a molecular genetic mechanism for the efficacy of Computerized Cognitive Remediation Therapy (CCRT) .

DETAILED DESCRIPTION:
Among the cognitive disorders of chronic schizophrenia, the most reported is the executive dysfunction of the prefrontal lobe. There is increasing evidence that Computerized Cognitive Remediation Therapy (CCRT) has a significant improvement in the implementation of schizophrenia, but the specific mechanism is unknown. Therefore, this study plans to select 154 patients with chronic schizophrenia who were hospitalized for a long time. They were randomly divided into two groups. The study group received antipsychotic drugs combined with Computerized Cognitive Remediation Therapy (CCRT) for 4 times/week for 45 minutes each time. The control group only received antipsychotic drugs. For a total of 12 weeks. brain-derived neurotrophic factor (BDNF) and tyrosine receptor kinase B(TRK-B) genes in peripheral blood were detected in both groups before and after treatment. Clinical symptoms and executive function assessment were performed in both groups before and after treatment. The relevance of genes and their effects on downstream protein expression levels led to a molecular genetic mechanism for the efficacy of Computerized Cognitive Remediation Therapy (CCRT).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years old, Han nationality, male or female;
2. Comply with the American Diagnostic Criteria for Mental Disorder (DSM-V) diagnostic criteria for "schizophrenia";
3. The course of the disease and continued treatment with antipsychotic drugs for > 2 years, stable for at least one month;
4. Positive NegativeSyndrome Scale (PANSS) < 70 points;
5. intelligence quotient (IQ)>80;
6. Cultural, social and educational backgrounds are sufficient to understand informed consent and research content.

Exclusion Criteria:

1. Concomitant diagnosis in addition to Diagnostic and Statistical Manual of Mental Disorders-V other than schizophrenia;
2. Central nervous system organic diseases;
3. There are alcohol or other substances dependent or abused in the past two months, causing significant social and cognitive impairment;
4. In the past year, there have been major life events such as widowhood;
5. Those who have serious suicide attempts (the third item of the (Hamilton Depression Scale-17,HAMD-17) scale "suicide" ≥ 3 points);
6. The current patient's severe unstable physical disease;
7. pregnant women and lactating women;
8. Those who have received modified electroconvulsive therapy (MECT) and repetitive Transcranial Magnetic Stimulation (rTMS) treatment in the past month;
9. Those who have been ineffective for more than 3 months of systemic psychotherapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The score of Positive and Negative Syndrome Scale (PANSS) | the baseline
  The score of Positive and Negative Syndrome Scale (PANSS) ranges from 19-133 and will be administered to assess the effectiveness of treatment. Do higher values represent a worse outcome. The subscales are summed to compute a total score.
The score of Positive and Negative Syndrome Scale (PANSS) | the end of 12 week
  The score of Positive and Negative Syndrome Scale (PANSS) ranges from 19-133 and will be administered to assess the effectiveness of treatment. Do higher values represent a worse outcome.The subscales are summed to compute a total score.
The concentration of Brain Derived Neurotrophic Factor (BDNF) used to assess the effectiveness of treatment | the baseline
  The Concentration of Brain Derived Neurotrophic Factor (BDNF) will be administered to assess the effectiveness of treatment. Do higher values represent a better outcome.
The concentration of Brain Derived Neurotrophic Factor (BDNF) used to assess the effectiveness of treatment | the end of 12 week
  The Concentration of Brain Derived Neurotrophic Factor (BDNF) will be administered to assess the effectiveness of treatment. Do higher values represent a better outcome.

SECONDARY OUTCOMES:
The concentration of tyrosine receptor kinase B(TRK-B) used to assess the effectiveness of treatment | the baseline
  The Concentration of tyrosine receptor kinase B(TRK-B) will be administered to assess the effectiveness of treatment. Do higher values represent a better outcome.
The concentration of tyrosine receptor kinase B(TRK-B) used to assess the effectiveness of treatment | the end of 12 week
  The Concentration of tyrosine receptor kinase B(TRK-B) will be administered to assess the effectiveness of treatment. Do higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: tao shen, professor, Study Director — Shanghai Huangpu District Health and Wellness Committee
Locations (1):
- Huangpu District Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03772951/Prot_SAP_ICF_001.pdf